CLINICAL TRIAL: NCT03778125
Title: Clinical and Microbiologic Outcomes in Patients Treated for Multidrug-resistant Shigella Infections in Dhaka, Bangladesh
Brief Title: Multidrug Resistant Shigella Infection in Bangladesh
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Virginia (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Eric R. Houpt, MD, Jack Gwaltney Professor of Infectious Diseases, University of Virginia
Other Study IDs: 21166; PR-18078 (Other: International Centre for Diarrhoeal Disease Research)
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Diarrhea; Shigella
Keywords: multidrug resistant
MeSH Terms: conditions — Diarrhea; Dysentery, Bacillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool culture positive for Shigella
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this project is to systematically collect clinical and nutritional outcomes information on patients treated for Shigella infection so that physicians and clinical laboratories can better define which Shigella infections are "resistant" to antibiotics and which are "susceptible", focusing on azithromycin a last-line drug to treat drug resistant Shigella

DETAILED DESCRIPTION:
2000 suspected Shigella cases will be recruited from International Centre for Diarrhoeal Disease Research hospital, Dhaka who are presenting with diarrhea at the hospital. A stool sample will be collected from the participants after consenting by the study staff. Stool microscopy will be performed to see the white blood cells(WBC) and red blood cells (RBC). If WBC > 10 HPF (4) with any RBC present, culture will be performed from this stool to identify Shigella. Such patients with invasive diarrhea are treated with azithromycin per local standard of care. Enrolled participant will be invited for further follow up when culture from the stool is Shigella positive. Minimal inhibitory concentration (MIC) testing of Shigella isolates and Molecular testing of Shigella isolates will be performed from Shigella cultures. This is an observational study. This study does not provide any treatment to the study participants; they will receive treatment as per International Centre for Diarrhoeal Disease Research Dhaka hospital guidelines. We will then examine the effect of the azithromycin minimal inhibitory concentration on clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* diarrheal illness less than 96 hours duration
* microscopic evidence of inflammatory diarrhea
* plus mucus in stool
* plus abdominal pain/cramps
* Subject or parents or legal guardian willing to come for follow up at hospital or allow study staff for home visit
* residence in Dhaka region
* presentation during daytime hours

Exclusion Criteria:

• Not receiving treatment with azithromycin at enrolment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 2000 suspected Shigella cases will be recruited from International Centre for Diarrhoeal Disease Research hospital, Dhaka who are presenting with diarrhea at the hospital. A stool sample will be collected from the participants after consenting by the study staff. Stool microscopy will be performed to see the white blood cells (WBC). If WBC > 10 HPF (4) culture will be performed from this stool to identify Shigella. Such patients with invasive diarrhea are treated with azithromycin per local standard of care. Enrolled participant will be invited for further follow up when culture from the stool is Shigella positive. Minimal inhibitory concentration (MIC) testing of Shigella isolates and Molecular testing of Shigella isolates will be performed from Shigella cultures.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome: resolution of diarrhea | Day 5
  resolution of diarrhea as measured by the participant through a memory aid

SECONDARY OUTCOMES:
Microbiologic outcome: Shigella negative cultures | Day 5
  Proportion shigella culture negative isolates
Proportion of patients that have complications | day 5
  required hospitalization or have extraintestinal complications

OTHER OUTCOMES:
time to last unformed stool | Day 5
  duration of diarrhea in days
fever | Day 5
  duration of fever in days
bloody stool | Day 5
  duration of bloody stool in days
difference in invasion plasmid antigen H (ipaH) | Day 5
  molecular detection of Shigella quantity

CONTACTS AND LOCATIONS:
Overall Officials: Eric R Houpt, MD, Principal Investigator — University of Virginia
Locations (1):
- International Centre for Diarrhoeal Disease Research, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Houpt ER, Ferdous T, Ara R, Ibrahim M, Alam MM, Kabir M, Platts-Mills J, Ahmed T, Faruque ASG, Taniuchi M, Haque R. Clinical Outcomes of Drug-resistant Shigellosis Treated With Azithromycin in Bangladesh. Clin Infect Dis. 2021 May 18;72(10):1793-1798. doi: 10.1093/cid/ciaa363. PMID 32239137